CLINICAL TRIAL: NCT04933617
Title: Phase 1 Study of Copanlisib With Dose-adjusted EPOCH-R in Relapsed and Refractory Burkitt Lymphoma and Other High-Grade B-cell Lymphomas
Brief Title: Copanlisib With Dose-Adjusted EPOCH-R in Relapsed and Refractory Burkitt Lymphoma and Other High-Grade B-cell Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early because copanlisib was removed from the market by the Food and Drug Administration (FDA) and the manufacturer.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000193; 000193-C
Record Dates: First submitted 2021-06-18; First posted 2021-06-22 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Burkitt Lymphoma; High-grade B-cell Lymphoma; T-cell/Histocyte-rich Large B-cell Lymphoma; Diffuse Large B-Cell Lymphoma (DLBCL); Germinal Center B-cell Type (GCB)
Keywords: Aliqopa; BAY 80-6946; Monoclonal Antibody; PI3K Target
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Etoposide; etoposide phosphate; copanlisib; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Echocardiography; Electrocardiography; Tomography, X-Ray Computed; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1- Dose Escalation, Original Copanlisib Intravenous (IV) (Experimental): Copanlisib intravenous (IV) per dose level (30 mg, 45 mg, or 60 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Interventions: Biological: Rituximab; Drug: Etoposide; Biological: Copanlisib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Diagnostic Test: ECHO; Diagnostic Test: EKG; Diagnostic Test: MRI Brain; Diagnostic Test: 18F-FDG - PET; Diagnostic Test: CT Scan; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Diagnostic Test: Lumbar Puncture (LP)
- Arm 2 - Dose Expansion, Modified Copanlisib Intravenous (IV) (Experimental): Copanlisib intravenous (IV) at the recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R). Up to 6 cycles total.
  Interventions: Biological: Rituximab; Drug: Etoposide; Biological: Copanlisib; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Diagnostic Test: ECHO; Diagnostic Test: EKG; Diagnostic Test: MRI Brain; Diagnostic Test: 18F-FDG - PET; Diagnostic Test: CT Scan; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Diagnostic Test: Lumbar Puncture (LP)

INTERVENTIONS:
Biological: Rituximab — Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Other Names: Rituxan
Drug: Etoposide — Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Other Names: Toposar; Etopophos
Biological: Copanlisib — Copanlisib intravenous (IV) is administered at a fixed dose (30 mg, 45 mg, or 60 mg) on days 1 and 5 of each 21-day cycle for up to 6 cycles
  Other Names: Aliqopa
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Other Names: Cytoxan
Drug: Doxorubicin — Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Other Names: Adriamycin
Drug: Vincristine — Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Other Names: Marqibo; Vincasar PFS
Drug: Prednisone — Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
  Other Names: Deltasone; Rayos; Prednisone Intensol
Diagnostic Test: ECHO — At screening.
  Other Names: Echocardiogram
Diagnostic Test: EKG — At screening.
  Other Names: Electrocardiogram
Diagnostic Test: MRI Brain — At screening.
  Other Names: Magnetic resonance imaging of the brain
Diagnostic Test: 18F-FDG - PET — At screening, baseline, after cycle 1, 3, and 6, and end of treatment.
  Other Names: Fludeoxyglucose F18
Diagnostic Test: CT Scan — At screening, baseline, after cycle 1, 3, and 6, end of treatment and follow-up.
  Other Names: Computed tomography scan
Procedure: Bone Marrow Aspiration — At screening and end of treatment.
Procedure: Bone Marrow Biopsy — At screening and end of treatment.
Diagnostic Test: Lumbar Puncture (LP) — Baseline and end of treatment.
  Other Names: Spinal tap

SUMMARY:
Background:

Burkitt Lymphoma (BL) and diffuse large B-cell lymphoma (DLBCL) are aggressive B cell lymphomas. Frontline treatment does not always work. Researchers want to see if a combination of drugs can help.

Objective:

To learn if it is safe to give people with certain cancers copanlisib together with rituximab and combination chemotherapy dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R).

Eligibility:

People ages 18 and older with relapsed and/or refractory highly aggressive B-cell lymphomas such as BL and certain types of diffuse large B-cell lymphoma (DLBCL).

Design:

Participants will be screened with:

Medical history

Physical exam

Bone marrow aspiration and biopsy. A needle will be put into their hipbone. Marrow will be removed.

Imaging scans of the chest, abdomen, pelvis, and/or brain

Tumor biopsy (if needed)

Blood and urine tests

Heart function tests

Treatment will be given in 21-day cycles for up to 6 cycles. Participants will get copanlisib by intravenous (IV) infusion. They will also get a group of medicines called DA-EPOCH-R, as follows. They will get rituximab by IV infusion. Doxorubicin, etoposide, and vincristine will be mixed together in an IV bag and given by continuous IV infusion over 4 days. They will get cyclophosphamide by IV infusion. They will take prednisone by mouth.

Participants will have frequent study visits. At these visits, they will repeat some screening tests. They may give tissue, saliva, and cheek swab samples. They will have at least one spinal tap. For this, a needle will be inserted into the spinal canal. Fluid will be removed.

Participants will have a visit 30 days after treatment ends. They will have follow-up visits for at least 5 years.

DETAILED DESCRIPTION:
Background:

Burkitt Lymphoma (BL) is a highly aggressive B cell lymphoma that often involves the bone marrow and central nervous system (CNS)

Frontline therapy cures 80-85% of adults with BL but patients with CNS involvement or those who relapse after frontline therapy are at high risk for treatment failure.

Diffuse large B-cell lymphoma (DLBCL) is a heterogeneous group of aggressive B-cell lymphomas that are successfully cured by frontline therapy in 60-70% of cases.

A subset of DLBCL that have myelocytomatosis (MYC) gene rearrangement as well as those that have transformed from an underlying indolent lymphoma have a lower cure rate.

Dose-adjusted dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) is an infusional chemotherapy platform often used as frontline therapy for these aggressive B-cell lymphomas and is an effective chemotherapy platform from which to rationally design novel therapies for patients with BL, high grade B-cell lymphomas-double hit/triple hit (HGBCL-DH/TH), DLBCL and myelocytomatosis (MYC) rearrangements, and other high-risk DLBCL

The phosphoinositide 3-kinase (PI3K) pathway is an important signaling pathway for cellular responses to growth factors and a downstream event of B-cell receptor signaling.

Copanlisib targets both PI3K-a and PI3K-d isoforms and is approved for relapsed follicular lymphoma (FL), active as monotherapy in DLBCL, and highly effective in pre-clinical models of BL.

Copanlisib crosses the blood brain barrier suggesting it may prevent secondary CNS spread in highly aggressive B-cell lymphomas.

Copanlisib is a rational targeted agent to be added to DA-EPOCH-R in patients with BL, HGBCL-DH/TH, and other high-risk B-cell lymphomas.

Objective:

To determine the Maximal tolerated dose (MTD) and Recommended Phase II dose (RP2D) of copanlisib in combination with DA-EPOCH-R in subjects with Burkitt lymphoma (BL) and high-grade B-cell lymphomas- double hit/triple hit (HGBCL-DH/TH) relapsed after or refractory to chemo-immunotherapy.

Eligibility:

Subjects must have a histologic diagnosis, confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) with one of the following subtypes and prior therapy, as follows:

Burkitt lymphoma, Burkitt-like lymphoma with 11q aberration, High-grade B-cell lymphoma, not otherwise specified (NOS), High-grade B-cell lymphoma, with MYC and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements - following at least 1 anthracycline-containing regimen.

OR

DLBCL, NOS, Germinal center B-cell type (GCB) type, T-cell/histocyte-rich large B-cell lymphoma, following at least 1 anthracycline-containing regimen AND at least 2 prior regimens OR be primary refractory to frontline therapy.

Age >= 18

Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Adequate bone marrow and organ function

Design:

Phase 1, open-label, single center, non-randomized

"3+3" dosing will be used to determine the recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of dose escalated copanlisib in combination with standard regimen DA-EPOCH-R

Maximum 6 cycles (21-day cycles) of combination therapy

Dose expansion at the RP2D or MTD to evaluate efficacy and further evaluate safety.

To explore all dose levels, including further evaluation in dose expansion cohort, the accrual ceiling will be set at 39.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must have a histologic diagnosis, confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) with one of the following subtypes and prior therapy, as follows:

  * At least 1 anthracycline-containing regimen:

    * Burkitt lymphoma
    * Burkitt-like lymphoma with 11q aberration
    * High-grade B-cell lymphoma, nor otherwise specified (NOS)
    * High-grade B-cell lymphoma, with myelocytomatosis (MYC) and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements

OR

--Must have had at least 2 prior regimens, 1 of which must have been anthracycline containing regimen OR be primary refractory to frontline therapy:

---Diffuse large B-cell lymphoma (DLBCL), NOS, Germinal center B-cell type (GCB) type;

NOTE: subjects with coexisting or a history of indolent lymphoma are eligible (i.e., transformed lymphoma)

---T-cell/histocyte-rich large B-cell lymphoma

* Measurable or evaluable disease on imaging scans or bone marrow
* No other current systemic anti-lymphoma therapy. NOTE: Recent short-term (less than or equal to 7 days) use of corticosteroids or prior radiation to sites of disease involvement is permitted.
* Any human immunodeficiency virus (HIV) status will be included in this study as long as infection is controlled; in the opinion of the investigator. Status must be confirmed at screening and the subject must be willing to take any recommended antiretroviral therapy.
* Greater than or equal to 18 years of age on day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ function as evidenced by the following laboratory parameters, unless dysfunction is secondary to lymphoma involvement as determined by the investigator:

  * Absolute neutrophil count (ANC) greater than or equal to 1,000/mm^3
  * Platelets greater than or equal to 100 x 10^9 /L
  * Hemoglobin greater than or equal to 8 g/dL (unless due to disease itself, transfusion permitted to meet criteria)
  * Renal function Glomerular filtration rate (GFR) greater than or equal to 50ml/min/1.73 m^2 as estimated by Modification of Diet in Renal Disease

Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, a 24- hour urine creatinine clearance can be used to directly measure.

* Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) OR < 1.5-3.0 x ULN for subjects with liver involvement*
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3.0 x ULN OR < 5 x ULN for subjects with liver involvement

  * Acceptable range, as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia.

    * Must have fully recovered from all effects of prior surgery. NOTE: Minor procedures requiring Twilight sedation, such as tissue biopsies, endoscopies or mediport placement require a 24-hour waiting period prior to treatment initiation.
    * Women of childbearing potential (WOCBP) and men with female partners of childbearing potential must agree to use a highly effective method of contraception when sexually active (intrauterine device, surgical sterilization, contraceptive rod, abstinence) for the time period between signing of the informed consent form and for at least 1 month after the last dose of copanlisib. WOCBP and men with female partners of childbearing potential must agree to use an effective method of contraception (two of the following: diaphragm, cervical cap, contraceptive sponge, condom, hormonal) when sexually active for the time period between signing of the informed consent and for at least 12 months after the last dose of rituximab. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.

NOTE: A woman is considered of childbearing potential, (i.e., fertile), following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the subject how to achieve highly effective birth control (failure rate of less than 1%), e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence.

* Willingness to have a central venous access line placed if the subject does not already have one in place
* Ability of patient to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Subjects previously exposed to, intolerant of, or ineligible for phosphoinositide 3-kinases (PI3K) inhibitors and/or their combination
* Brain parenchymal involvement
* Patients who have been treated with prior chimeric antigen receptor (CAR)-T therapy or any regimen containing fludarabine.
* Cytomegalovirus (CMV)-positive polymerase chain reaction (PCR) at screening
* History of diabetic ketoacidosis
* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the subject at the discretion of the investigator:

  * Any secondary malignancy that requires active systemic therapy
  * Diabetes mellitus with hemoglobin (Hgb) hemoglobin A1C (A1C) > 8.5
  * Clinically significant interstitial lung disease and/or lung disease that severely impairs lung function
  * Uncontrolled human immunodeficiency virus (HIV)
  * Active hepatitis C infection. NOTE: Subjects who are hepatitis C antibody positive will need to have a negative hepatitis C virus (HCV) PCR result before enrollment. Those with a positive PCR for hepatitis C are excluded.
  * Active hepatitis B infection. NOTE: Patients who are hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) positive will need to have a negative HBV PCR result before enrollment. Those with a positive PCR for hepatitis B are excluded. Those who are hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) positive with a negative PCR for hepatitis B will be treated with antivirals designed to prevent hepatitis B reactivation (e.g., entecavir) throughout therapy and for 12 months after therapy and have monitoring for hepatitis B reactivation with PCR.
  * Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
    * Congestive heart failure (New York Heart Association functional classification III-IV)
    * Unstable angina
    * Left Ventricular Ejection Fraction (LVEF) <40% as determined by echocardiogram (ECHO) at screening
    * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II and third-degree AV block)
    * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

      * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
      * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
      * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
  * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the subject inappropriate for entry into the study.
* Requirement to continue on any of the medications that are excluded
* Breast-feeding subjects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All large- scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000193-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous 30mg intravenous (IV) on days 1 and 5 of each 21-day cycle for up to 6 cycles
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
- Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous 30mg intravenous (IV) on day 1 of each 21-day cycle for up to 6 cycles
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
- Dose Escalation: Arm 1, Dose Level 2, Original: 45mg Copanlisib: Copanlisib intravenous (IV) per dose level (45 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous 45mg intravenous (IV) on day 1 of each 21-day cycle for up to 6 cycles
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
- Dose Escalation: Arm 1, Dose Level 1, Modified: 60mg Copanlisib: Copanlisib intravenous (IV) per dose level (60 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous 60mg intravenous (IV) on day 1 of each 21-day cycle for up to 6 cycles
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
- Arm 2 - Dose Expansion, Modified Copanlisib: Copanlisib intravenous (IV) at the recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R). Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg, 45 mg, or 60 mg) on day 1 of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
Period: Dose Escalation
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 2, Original: 45mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 60mg Copanlisib | Arm 2 - Dose Expansion, Modified Copanlisib
Started | 5 | 3 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0
Not completed — Early closure of study | 0 | 3 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 2, Original: 45mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 60mg Copanlisib | Arm 2 - Dose Expansion, Modified Copanlisib
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on days 1 and 5 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg) on days 1 and 5 of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
- Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg) on day 1 of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 44 [22 to 59] | 43 [36 to 82] | 43.5 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D)
Description: MTD and RP2D is defined as the dose level at which no more than 1 of up to 6 participants experience dose limiting toxicity (DLT) during the DLT period, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of treatment. A DLT is any treatment-emergent, clinically relevant, and related severe (grade ≥ 3) toxicity that is possibly, probably, or definitely related to copanlisib.
Time Frame: 21 days
Measure: Number; unit: Mg
Groups:
- All Participants: All participants treated with 30mg copanlisib in dose level 1.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Mg | NA — Due to early termination of the study, a maximum tolerated dose or recommended phase 2 dose could not be assessed. Additional participants were required to assess the recommended phase 2 dose.

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is the best response recorded from the start of the treatment until disease progression/recurrence determined by Kaplan-Meier method and reported along with a 95% confidence interval. Response was assessed by the Revised Response Criteria for Malignant Lymphoma criteria, and the Lugano Classification Response Criteria for Non-Hodgkin Lymphoma (NHL). Complete response (CR) is complete disappearance of all detectable evidence of disease and disease-related symptoms. Partial response (PR) is a ≥50% decrease in the sum of the product of the diameters of up to 6 of the largest dominant nodes or nodal masses. Progressive disease (PD) is appearance of any new nodal lesion ≥1.6 cm in greatest tumor dimension or ≥1.1 cm in short axis during or after the end of therapy. A participant is considered to have stable disease (SD) when he or she fails to attain the criteria needed for a CR, PR, or Minimal Response (MR) but does not fulfill those for PD.
Time Frame: Response was assessed after cycles 1, 3 and 6 (each cycle is 21 days), approximately 63 days.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg) on day 1 of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Percentage of participants
  Complete Response | 0 [0 to 52.2] | 66.7 [9.4 to 99.2]
  Partial Response | 40 [5.3 to 85.3] | 33.3 [0.8 to 90.6]
  Progressive Disease | 20 [0.5 to 71.6] | 0 [0 to 70.8]
  Stable Disease | 40 [5.3 to 85.3] | 0 [0 to 70.8]
  Minimal Response | 0 [0 to 52.2] | 0 [0 to 70.8]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first, assessed every 3-6 months The progression free survival will be determined by the Kaplan-Meier method and reported along with a 95% confidence interval. Response was assessed by the Revised Response Criteria for Malignant Lymphoma criteria, and the Lugano Classification Response Criteria for Non-Hodgkin Lymphoma (NHL). Disease relapse is Progressive disease (PD) is appearance of any new nodal lesion ≥1.6 cm in greatest tumor dimension or ≥1.1 cm in short axis during or after the end of therapy or increase by ≥50% from PPD (cross product of the longest transverse diameter and perpendicular diameter) nadir.
Time Frame: Time from enrollment to progression or death, approximately 9 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Months | 3.0 [0.5 to 6.3] | 5.4 [NA to NA] — There is only one observation out far enough to be used to compute the median, and thus there is no way to get an estimate of the variability of the median.

4. Secondary Outcome: Complete Response Rate
Description: Response was assessed by the Revised Response Criteria for Malignant Lymphoma criteria, and the Lugano Classification Response Criteria for Non-Hodgkin Lymphoma (NHL). Complete response (CR) is complete disappearance of all detectable evidence of disease and disease-related symptoms. The response rate will be determined by Kaplan-Meier method and reported along with a 95% confidence interval.
Time Frame: Response was assessed after cycles 1, 3 and 6 (each cycle is 21 days). Approximately 63 days.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Percentage of participants | 0 [0 to 52.2] | 66.7 [9.4 to 99.2]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of study enrollment until death from any cause, assessed every 3-6 months. OS will be determined by the Kaplan-Meier method and reported along with a 95% confidence interval.
Time Frame: Time from enrollment to death, approximately 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Months | 5.9 [0.5 to 7.6] | NA [NA to NA] — OS is undefined because none of the participants died by the end of follow-up

6. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the time from the date of study enrollment until time of disease relapse from complete response (CR), disease progression, initiation of subsequent systemic anti-lymphoma therapy for either positron-emission tomography (PET)-positive or biopsy-proven residual disease, or death, whichever occurs first. The EFS will be determined by the Kaplan-Meier method and reported along with a 95% confidence interval. Response was assessed by the Revised Response Criteria for Malignant Lymphoma criteria, and the Lugano Classification Response Criteria for Non-Hodgkin Lymphoma (NHL). Complete response (CR) is complete disappearance of all detectable evidence of disease and disease-related symptoms. Progressive disease (PD) is appearance of any new nodal lesion ≥1.6 cm in greatest tumor dimension or ≥1.1 cm in short axis during or after the end of therapy. Disease relapse is Progressive disease (PD), an appearance of any new nodal lesion ≥1.6 cm in greatest tumor dimension.
Time Frame: Time from enrollment to next line of anti-lymphoma therapy, progressive disease, or death. Approximately 6 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Months | 1.9 [0.5 to 3.0] | 5.4 [NA to NA] — There is only one observation out far enough to be used to compute the median, and thus there is no way to get an estimate of the variability of the median.

7. Secondary Outcome: Number of Serious and/or Non-serious Grades 3-5 Adverse Events Related to Copanlisib
Description: Rate and severity of adverse events (AEs) summarized by grade and type of toxicity. AE's were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: An average of 245.5 days
Measure: Number; unit: Adverse events
Groups:
- Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on day 1 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg) on day of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Adverse events
  Grade 3 Serious Febrile Neutropenia | 1 | 0
  Grade 3 Serious Generalized muscle weakness | 1 | 0
  Grade 4 Serious Febrile Neutropenia | 1 | 0
  Grade 4 Serious Platelet Count Decreased | 1 | 0
  Grade 5 Serious Multi-organ Failure | 1 | 0
  Grade 3 Non-serious Anemia | 2 | 0
  Grade 3 Non-serious Hyperglycemia | 1 | 0
  Grade 3 Non-serious Platelet Count Decreased | 1 | 2
  Grade 3 Non-serious Neutrophil Count Decreased | 0 | 1
  Grade 4 Non-serious Neutrophil Count Decreased | 1 | 2
  Grade 4 Non-serious Platelet Count Decreased | 5 | 1

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 245.5 days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib: Copanlisib intravenous (IV) per dose level (30 mg) on days 1 and 5 of each 21-day cycle in combination with standard dosing dose adjusted rituximab, etoposide, prednisolone, vincristine, cyclophosphamide, doxorubicin (DA-EPOCH-R) to determine recommended phase 2 dose (RP2D) and maximum tolerated dose (MTD) of copanlisib. Up to 6 cycles total.
  Rituximab: Rituximab 375 mg/m^2 intravenous (IV) per protocol on Day 1 of each cycle up to 6 cycles
  Etoposide: Etoposide 50 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Copanlisib: Copanlisib intravenous (IV) is administered at a fixed dose (30 mg) on day 1 of each 21-day cycle for up to 6 cycles.
  Cyclophosphamide: Cyclophosphamide 750 mg/m^2 intravenous (IV) on Day 5 of each cycle up to 6 cycles
  Doxorubicin: Doxorubicin 10 mg/m^2/day continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Vincristine: Vincristine 0.4 mg/m^2/day (no cap) continuous intravenous infusion (CIVI) on Days 1-4 of each cycle up to 6 cycles
  Prednisone: Prednisone 60 mg/m^2 by mouth (PO) twice a day (BID) Days 1-5 (total 120mg/m^2/day)
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Participants | 5 | 3

9. Other Pre Specified Outcome: Number of Participants With Dose Limiting-toxicity (DLT)
Description: A DLT is any treatment-emergent, clinically relevant, and related severe (grade ≥ 3) toxicity that is possibly, probably or definitely related to copanlisib.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
Number analyzed (Participants) | 5 | 3
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 245.5 days.
Arm/Group | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib
All-Cause Mortality (participants affected / at risk) | 5/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib (N=5) | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: Arm 1, Dose Level 1, Original: 30mg Copanlisib (N=5) | Dose Escalation: Arm 1, Dose Level 1, Modified: 30mg Copanlisib (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (8) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (3)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 3 (7) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04933617/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Screening Affected Subject Consent (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04933617/ICF_001.pdf
  • Informed Consent Form: Cohort Standard Affected Subject Consent (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04933617/ICF_002.pdf